CLINICAL TRIAL: NCT05345002
Title: A Phase 2 Trial of All-Trans Retinoic Acid (ATRA) Plus PD-1 Inhibition in Recurrent IDH-Mutant Glioma
Brief Title: All-Trans Retinoic Acid (ATRA) Plus PD-1 Inhibition in Recurrent IDH-Mutant Glioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stephen Bagley, MD, MSCE (Other)
Collaborators: Incyte Corporation (Industry); Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor-Investigator, Stephen Bagley, MD, MSCE, Assistant Professor of Medicine, Abramson Cancer Center at Penn Medicine
Organization: Abramson Cancer Center at Penn Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 02322
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Glioma; IDH Mutation; Astrocytoma; Oligodendroglioma
MeSH Terms: conditions — Glioma; Astrocytoma; Oligodendroglioma | interventions — Tretinoin

STUDY DESIGN:
Intervention Model Description: The study has a Safety Run-In, a Phase 2 Portion with Arm A and Arm B and a Surgical Portion with Arm C and Arm D. .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A (failed prior TMZ + one other alkylating chemotherapy) (Experimental): Subjects in Arm A are alkylator-refractory and at high risk for progression of disease, have failed temozolmide and another alkylating agent. Subjects in Arm A will receive 28-day cycles of treatment, with ATRA 45mg/m2/day given orally in two equally divided doses on days 1 through 14 and retifanlimab 500mg IV on day 1.
  Interventions: Drug: Retifanlimab; Drug: All-trans retinoic acid
- Arm B (failed only one prior alkylating chemotherapy) (Experimental): Subject in Arm B are patients who have failed only one prior alkylating chemotherapy regimen and have gone at least 12 months since the last treatment. Subjects in Arm B will receive 28-day cycles of treatment, with ATRA 45mg/m2/day given orally in two equally divided doses on days 1 through 14 and retifanlimab 500mg IV on day 1.
  Interventions: Drug: Retifanlimab; Drug: All-trans retinoic acid
- Arm C (surgical arm, ATRA alone pre-operatively) (Experimental): Subject in Arm C will receive ATRA 45mg/m2/day orally in two equally divided doses for 14 days pre-surgery, then undergo surgery. Following surgery all patients will receive 28-day cycles of treatment, with ATRA 45mg/m2/day given orally in two equally divided doses on days 1-14 and retifanlimab 500mg IV on day 1.
  Interventions: Drug: Retifanlimab; Drug: All-trans retinoic acid
- Arm D (surgical arm, ATRA + retifanlimab pre-operatively) (Experimental): Subject in Arm D will receive the combination of ATRA 45mg/m2/day orally in two equally divided doses for 14 days pre-surgery plus a 500mg IV dose of retifanlimab 14 days prior to the date of surgery. Following surgery all patients will receive 28-day cycles of treatment, with ATRA 45mg/m2/day given orally in two equally divided doses on days 1-14 and retifanlimab 500mg IV on day 1.
  Interventions: Drug: Retifanlimab; Drug: All-trans retinoic acid

INTERVENTIONS:
Drug: Retifanlimab — Administered 500mg IV on day 1 of every 28-day cycle, continued until disease progression, unacceptable toxicity, or 2 years from the first dose of study medication, whichever occurs first.
Drug: All-trans retinoic acid — All-trans retinoic acid (ATRA) 45mg/m2 orally in two equally divided doses on days 1-14 of each 28-day cycle, continued until disease progression, unacceptable toxicity, or 2 years from the first dose of study medication, whichever occurs first.

SUMMARY:
This is a Phase II study of the combination of All-Trans Retinonic Acid (ATRA) and PD-1 inhibition (Retifanlimab) in patient with recurrent IDH-mutant glioma. The Sponsor-Investigator hypothesizes that the proposed regimen will be safe and stimulate a robust anti-tumor immune response.

DETAILED DESCRIPTION:
The study has a Safety Run-In, a Phase 2 Portion, and a Surgical Portion. The Phase 2 portion and Surgical portion will open to enrollment simultaneously following successful completion of the Safety Run-In.

Safety Run-In subjects receive 28-day cycles of treatment, with ATRA 45mg/m2/day given orally in two equally divided doses on days 1-14 and retifanlimab 500mg IV on day 1. Once Safety Run-In is complete, the Phase 2 and Surgical cohorts will commence uninterrupted.

Phase 2: All Phase 2 patients will receive 28-day cycles of treatment, with ATRA 45mg/m2/day given orally in two equally divided doses on days 1 through 14 and retifanlimab 500mg IV on day 1.

Arm A includes alkylator-refractory patients at high risk for progression of disease, having failed temozolomide and another alkylating agent. At the first stage, 12 subjects will be enrolled onto the study. This arm of the trial will be stopped if no response was obtained among the first 12 subjects (0/12). Otherwise, this arm of the study will continue to stage Four additional subjects will be enrolled on the second stage of this arm of the trial.

Arm B includes patients who have failed only one prior alkylating chemotherapy regimen and have gone at least 12 months since the last treatment (chemotherapy or radiation therapy), i.e., favorable risk patients. At the first stage, 14 subjects will be enrolled onto the study. This arm of the trial will be stopped if 5 or fewer responses were obtained among the first 14 subjects greater than or equal to 5 out of 14 subjects. Otherwise, this arm of the study will continue to stage 2. Three additional subjects will be enrolled on the second stage of this arm of the trial.

Surgical Portion: This portion of the study will enroll patients who are eligible for re-resection at the time of recurrence. Prior to surgical resection, patients are randomized 1:1 to receive either 1) single-agent ATRA 45mg/m2/day orally in two equally divided doses for 14 days pre-surgery (Arm C), or 2) the combination of ATRA 45mg/m2/day orally in two equally divided doses for 14 days pre-surgery plus a 500mg IV dose of retifanlimab 14 (+/-3) days prior to the date of surgery (Arm D). At surgery fresh tumor tissue will be collected for correlative studies. Following surgery all patients will receive 28-day cycles of treatment, with ATRA 45mg/m2/day given orally in two equally divided doses on days 1-14 and retifanlimab 500mg IV on day 1.

ELIGIBILITY:
Inclusion Criteria:

1. Prior histopathologically proven diagnosis of astrocytoma (grade 2-4) or oligodendroglioma (grade 2-3) according to the World Health Organization (WHO) 2021 Classification System that is progressive or recurrent following at least one prior alkylating chemotherapy regimen (i.e., temozolomide and/or lomustine), +/- radiation therapy
2. Patient's tumor must have a known mutation in IDH1 or IDH2. IDH1/2 mutation status must be confirmed by DNA sequencing and could have been performed in any CLIA/CAP-certified laboratory. IDH1/2 mutational testing could have been performed on patient's tumor either at initial diagnosis or on a subsequent recurrent tumor.
3. Safety Run-In and Phase 2 (Arm A and Arm B) patients:

   * All Safety Run-In and Phase 2 patients: patients with any contrast-enhancing tumor must have measurable disease per RANO criteria (defined by at least 1cmx1cm of contrast-enhancing tumor). Patients with exclusively non-enhancing tumors must have least a 25% increase in bi-dimensional product of FLAIR signal abnormality (measurable disease) compared to the patient's best MRI scan (smallest bi-dimensional product of FLAIR signal abnormality) obtained following completion of the patient's most recent line of therapy
   * Safety Run-In: Must have failed temozolomide OR another alkylator (e.g. lomustine, procarbazine, carmustine). May have failed an unlimited number of prior systemic regimens, +/- prior radiotherapy.
   * Arm A: Must have failed temozolomide AND another alkylator (e.g. lomustine, procarbazine, carmustine). May have failed an unlimited number of prior systemic regimens, +/- prior radiotherapy.
   * Arm B: Must have failed temozolomide OR another alkylator (maximum one prior chemotherapy regimen) +/- prior radiotherapy, AND must have gone at least 12 months since last treatment (chemotherapy or radiotherapy).
4. Surgical patients (Arm C and Arm D):

   * Must have clinical indication for surgical resection of the suspected recurrent/progressive tumor, as determined by patient's care providers; measurable disease is not required
   * 5-aminolevulinic acid (5-ALA) is not allowed for intraoperative tumor visualization due to the photosensitizing agent interaction with ATRA
   * Patient may have had an unlimited number of relapses and prior therapy regimens
5. Patient must have documented 1p/19q and O-6-methylguanine-deoxyribonucleic acid (DNA) methyltransferase (MGMT) methylation testing. If either of these has not been performed previously, they can be done prior to enrollment.
6. Patients must be able to undergo MRI of the brain with gadolinium. Patients must be maintained on a stable or decreased dose of corticosteroid regimen (no increase for 5 days) prior to this baseline MRI.
7. Patients must have recovered from severe toxicity of prior therapy; the following intervals from previous treatments are required to be eligible:

   * 12 weeks from completion of radiation
   * 6 weeks from a nitrosourea cytotoxic chemotherapy
   * 3 weeks from a non-nitrosourea cytotoxic chemotherapy
   * 4 weeks from any investigational (not Food and Drug Administration [FDA]-approved) agents, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter
   * 2 weeks from administration of a non-cytotoxic, FDA-approved agent (e.g. abemaciclib, olaparib, etc)
8. If patient is on systemic corticosteroids to treat brain edema and/or brain edema-related symptoms, the dose must be 2mg of dexamethasone (or equivalent) daily or less for a minimum of 5 days prior to first dose of retifanlimab.
9. Patients must be able to swallow oral medications
10. Age 18 or older
11. Karnofsky performance status greater than or equal to 60
12. Life expectancy >3 months
13. Adequate organ and marrow function:

    * Total bilirubin <1.5 x upper limit of normal (ULN) (except patients with suspected Gilbert's Syndrome, who are eligible for the study but exempt from the total bilirubin eligibility criterion)
    * ALT and AST ≤ 2.5x ULN
    * Calculated CrCl ≥ 30 ml/min (glomerular filtration rate can also be used in place of CrCl)
    * Absolute Neutrophil count ≥1,500/uL
    * Platelets ≥ 100,000/uL
    * Hemoglobin ≥ 9 g/dL
14. Reproductive Status

    1. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to the start of study drug.
    2. b) Women must agree to not breastfeed during the study or for 180 days after the last dose of study treatment
    3. WOCBP must agree to use an adequate method to avoid pregnancy (as defined below) from the time of study screening through 180 days from last dose of study drug
    4. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception (as defined below) starting with the first dose of study drug through 180 days after the last dose of study
    5. Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, these WOCBP must still undergo pregnancy testing as described in this section.

    At a minimum, participants of childbearing potential who are sexually active and their partners must agree to the use of a highly effective form of contraception (as defined below) throughout their participation beginning with the time of consent, during the study treatment, and for 180 days after last dose of study treatment(s).

    HIGHLY EFFECTIVE METHODS OF CONTRACEPTION:
    * Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants and intrauterine devices (IUDs) by WOCBP subject or male subject's WOCBP partner. Female partners of male subjects participating in the study may use hormone-based contraceptives as one of the acceptable methods of contraception since they will not be receiving study drug
    * Nonhormonal IUDs
    * Bilateral Tubal ligation
    * Vasectomy
    * Sexual Abstinence

      * It is not necessary to use any other method of contraception when complete abstinence is elected.
      * WOCBP participants who choose complete abstinence must continue to have pregnancy tests.
      * Acceptable alternate methods of highly effective contraception must be discussed in the event that the WOCBP participants chooses to forego complete abstinence.
15. Participant must, in the opinion of the Investigator, be able to comply with study procedures
16. Patients must be able to understand the study procedures and agree to participate in the study by providing written informed consent (or have legally authorized representative sign on patient's behalf if patient physically unable to sign consent due to neurologic deficit)

Exclusion Criteria:

Any of the following would exclude the subject from participation in the study:

1. Contrast-enhancing tumor in brainstem or spinal cord (subjects do not need spinal MRI for screening, but known spinal cord tumor is exclusionary)
2. Diffuse leptomeningeal disease
3. Patients who have received bevacizumab within the last 3 months are ineligible
4. Patients with clinically significant mass effect or midline shift (e.g., 1-2 cm of midline shift)
5. Use of any immunosuppressive medication other than steroids, including but not limited to antimetabolites, calcineurin inhibitors, and/or anti-TNF agents within six months of start of study drug
6. Prior diagnosis of immunodeficiency
7. Prior solid organ or bone marrow transplantation
8. Active autoimmune disease requiring systemic immunosuppression in excess of physiologic maintenance doses of corticosteroids (> 10 mg/day of prednisone or equivalent).

   * Physiologic corticosteroid replacement therapy at doses ≤ 10 mg/day of prednisone or equivalent for adrenal or pituitary insufficiency and in the absence of active autoimmune disease is permitted.
   * Participants with asthma that requires intermittent use of bronchodilators, inhaled corticosteroids, or local corticosteroid injections may participate.
   * Participants using topical, ocular, intra-articular, or intranasal corticosteroids (with minimal systemic absorption) may participate.
   * Brief courses of corticosteroids for prophylaxis (eg, contrast dye allergy) or study treatment-related standard premedications are permitted.

   EXCEPTIONS: Patients with the following autoimmune diseases may participate: type I diabetes mellitus, hypothyroidism only requiring hormone replacement, Grave's disease that is previously treated with thyroidectomy or radioiodine, celiac disease with symptoms controlled with a gluten-free diet.
9. Evidence of interstitial lung disease, history of interstitial lung disease, or active, noninfectious pneumonitis.
10. Immune related toxicity during prior checkpoint inhibitor therapy for which permanent discontinuation of therapy was recommended (per product label or consensus guidelines) or any immune-related toxicity requiring intensive or prolonged immunosuppression to manage (with the exception of endocrinopathy that is well controlled on replacement hormones).
11. Known active hepatitis B virus (HBsAg reactive) or active hepatitis C virus (HCV RNA detectable by PCR)
12. Human immunodeficiency virus (HIV)-positive patients on antiretroviral therapy
13. Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen are excluded from this trial. Otherwise, patients with prior or concurrent malignancy are eligible.
14. Any serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection that, in the opinion of the investigator, would put the subject at undue risk from the study treatment.
15. Patients with uncontrolled or significant cardiovascular disease including, but not limited to, any of the following are ineligible:

    * Myocardial infarction or uncontrolled angina within 90 days prior to consent
    * History of clinically significant arrhythmia (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
    * History of cardiomyopathy, pericarditis, significant pericardial effusion, myocarditis, or New York Heart Association (NYHA) functional class III-IV congestive heart failure
16. Known hypersensitivity to another monoclonal antibody that cannot be controlled with standard measures (e.g., antihistamines and corticosteroids)
17. Known allergy or hypersensitivity to any component of retifanlimab or formulation components.
18. Known allergy or hypersensitivity to all-trans retinoic acid (tretinoin), any of its components, or other retinoids
19. Prisoners or subjects who are involuntarily incarcerated
20. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness
21. Pregnant women are excluded
22. Has received a live vaccine within 28 days before the planned start of study treatment

    Note: Examples of live vaccines include but are not limited to measles, mumps, rubella, varicella-zoster (chickenpox), yellow fever, rabies, BCG, and typhoid vaccines. Seasonal influenza vaccines for injection are generally killed-virus vaccines and are allowed; however, intranasal influenza vaccines are live, attenuated vaccines and are not allowed.
23. Participant must not be simultaneously enrolled in any interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective radiographic response (ORR) | 26 months
  Objective radiographic response (ORR), as measured by modified Response Assessment in Neuro-Oncology (RANO) criteria. ). The response is classified as Complete Response (CR), Partial Response (PR), Stable Disease (SD), and Progressive Disease (PD).

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by NCI CTCAE v 5.0 | 25 months
  Adverse events will be evaluated by monitoring frequency, duration, and severity of adverse events (AEs) per NCI CTCAE v 5.0
Progression Free Survival | 84 months
  PFS, defined as the time from date of enrollment until the earliest date of disease progression (as determined by modified RANO criteria) or death due to any cause
Overall survival | 84 months
  OS, defined as the time from date of enrollment until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bagley, MD MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No